CLINICAL TRIAL: NCT05347667
Title: Influence of Menstrual Cycle Phase and Oral Contraceptive Pill (OCP) Use on the Muscle Protein Synthetic Response to Exercise in Young, Healthy Women
Brief Title: Menstrual Cycle Phase and Oral Contraceptive Pill (OCP) Use on Muscle Protein Synthesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Natural Science and Engineering Research Council of Canada (NSERC) (Unknown)
Responsible Party: Principal Investigator, Stuart Phillips, Professor, McMaster University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 14067
Record Dates: First submitted 2022-04-21; First posted 2022-04-26 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-12

CONDITIONS: Menstrual Cycle; Resistance Exercise; Muscle Protein Synthesis; OCP

STUDY DESIGN:
Intervention Model Description: In a randomized fashion, participants will have one leg undergo unilateral resistance exercise training to assess the muscle protein synthetic response in each menstrual cycle phase OR each pill phase (active vs. placebo)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre-Ovulation Unilateral Resistance Exercise OR Active OCP Phase (Experimental): One leg will undergo 2 sessions of unilateral resistance exercise during the follicular phase of the menstrual cycle (pre-ovulation) OR during the active phase of taking the OCP
  Interventions: Other: Unilateral Resistance Exercise Leg; Other: Control Leg
- Post-Ovulation Unilateral Resistance Exercise OR Inactive OCP Phase (Experimental): One leg will undergo 2 sessions of unilateral resistance exercise during the luteal phase of the menstrual cycle (post-ovulation) OR during the inactive phase of taking the OCP
  Interventions: Other: Unilateral Resistance Exercise Leg; Other: Control Leg

INTERVENTIONS:
Other: Unilateral Resistance Exercise Leg — One leg will perform unilateral resistance exercise
Other: Control Leg — One leg will serve as a non-exercise control

SUMMARY:
Skeletal muscle size and function is regulated by various factors, including hormones. While we understand the role of male sex hormones (testosterone), we aren't sure how female sex hormones (estrogen and progesterone) influence muscle mass and strength. Female physiology is unique in that hormones fluctuate throughout the menstrual cycle. In the first phase (follicular phase) following menstruation, estrogen levels are high while progesterone levels are low. In the second phase (luteal phase), progesterone levels are high. Females are often excluded from studies because researchers are concerned that the menstrual cycle might affect the results. The purpose of this study is to investigate the response to resistance exercise in each phase of the menstrual cycle.

ELIGIBILITY:
Inclusion Criteria:

* Healthy females, between the ages of 18 and 30 y with a regular menstrual cycle
* Body Mass Index between 18.5 and 30.0 kg/m2
* Able and willing to provide informed consent

Exclusion Criteria:

* A history of neuromuscular disorders or muscle/bone wasting diseases
* Any acute or chronic illness, cardiac, pulmonary, liver, or kidney abnormalities, uncontrolled hypertension, insulin-dependent or insulin-independent diabetes, or the presence of any other metabolic disease - all of which will be determined via a medical history screening questionnaire
* The use of any medications known to affect protein metabolism (glucocorticoids, non-steroidal anti-inflammatory medication, or prescription strength acne medication, etc.)
* A (family) history of thrombosis
* The use of anticoagulant medications
* Consumption of tobacco-containing products
* Excessive alcohol consumption (>21 units/wk)
* History of bleeding diathesis, platelet or coagulation disorders
* Currently pregnant
* Irregular menstrual cycle as defined in the study protocol

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Change in Rates of Muscle Protein Synthesis | 6 days
  The investigators will use deuterated water and skeletal muscle biopsies to calculate the synthesis of skeletal muscle proteins.

SECONDARY OUTCOMES:
Whole-body proteolysis | 6 days
  The investigators will use 3-methylhistidine in urine to calculate the rate of whole-body myofibrillar protelysis

CONTACTS AND LOCATIONS:
Locations (1):
- Exercise Metabolism Research Laboratory, McMaster Univeristy, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
All participants will be assigned a unique subject ID, and therefore, other researchers involved with analyses will not have access to identifying participant information.

REFERENCES:
- [Result] Colenso-Semple LM, McKendry J, Lim C, Atherton PJ, Wilkinson DJ, Smith K, Phillips SM. Menstrual cycle phase does not influence muscle protein synthesis or whole-body myofibrillar proteolysis in response to resistance exercise. J Physiol. 2025 Mar;603(5):1109-1121. doi: 10.1113/JP287342. Epub 2024 Dec 4. PMID 39630025